CLINICAL TRIAL: NCT00888381
Title: A Phase IV, Single-centre, Open-label Study to Evaluate the Immunogenicity and Safety of the 2009/2010 Formulation of the Enzira® Vaccine in Two Groups of Healthy Volunteers: 'Adults' (Aged ≥ 18 to < 60 Years) and 'Older Adults' (Aged ≥ 60 Years).
Brief Title: A Study to Assess the Immunogenicity and Safety of CSL's 2009 / 2010 Formulation of Enzira® Vaccine in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSLCT-NHF-09-57; 2009-011450-18 (EudraCT Number)
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Adults (Experimental): Healthy volunteers aged 18 to 59 years
  Interventions: Biological: Inactivated Influenza Vaccine (2009 / 2010 formulation)
- Older Adults (Experimental): Healthy volunteers aged 60 years or older
  Interventions: Biological: Inactivated Influenza Vaccine (2009 / 2010 formulation)

INTERVENTIONS:
Biological: Inactivated Influenza Vaccine (2009 / 2010 formulation) — A single 0.5mL intramuscular injection into the deltoid region of the arm on Day 0.
  Other Names: Enzira® vaccine (2009 / 2010 formulation)

SUMMARY:
The purpose of the study is to assess the efficacy and safety of CSL's 2009/2010 formulation of the Enzira vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 years at the time of providing informed consent
* Participants are capable of understanding the purposes and risks of the study and are able to provide written informed consent
* Willing and able to adhere to all protocol requirements
* Able to provide a sample of approximately 17 mL of venous blood on two separate occasions without undue distress/discomfort
* Females of child bearing potential (i.e. ovulating, pre-menopausal, not surgically sterile) must be abstinent or be willing to use a medically accepted contraceptive regimen for the duration of the study

Exclusion Criteria:

* Known hypersensitivity to a previous dose of influenza vaccine or allergy to eggs, chicken protein, neomycin, polymyxin, or any components of the Enzira® vaccine
* Clinical signs of an active infection and/or an elevated oral temperature (≥ 38.0°C) at study entry
* A clinically significant medical or psychiatric condition
* A confirmed or suspected immunosuppressive condition
* History of seizures
* History of Guillain-Barré Syndrome
* Vaccination with a seasonal influenza virus vaccine or with an experimental influenza virus vaccine in the 6 months preceding study entry
* Currently receiving treatment with radiotherapy or cytotoxic drugs, or have received such treatment within the 6 months preceding administration of Enzira® vaccine
* Currently receiving systemic glucocorticoid therapy (excluding topical or inhaled preparations) or have received such therapy within the 3 months preceding study entry
* Currently receiving immunoglobulins and/or any blood products or have received such treatment within the 3 months preceding the administration of Enzira® vaccine
* Currently participating in another investigational study or recent study participation ending 3 months preceding administration of Enzira® vaccine
* Currently receiving treatment with warfarin or other anticoagulants
* Evidence or history of substance or alcohol abuse within the 12 months before study entry
* Females of child bearing potential who are planning to become pregnant or planning to discontinue contraceptive precautions during the study period
* Females who are pregnant or lactating
* Any issues that, in the opinion of the investigator, would render the subject unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director Vaccines, Study Director — Seqirus
Locations (1):
- Chiltern (Early Phase) Limited. Ninewells Hospital and Medical School, Dundee, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adults | Older Adults
Started | 60 | 60
Completed | 60 | 59
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults | Older Adults | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (12.31) | 66.2 (5.92) | 50.7 (18.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 56
  Male | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Evaluable Participants Achieving Seroconversion or Significant Increase in Antibody Titre.
Description: As per the criteria specified in the CPMP/BWP/214/96 Note for Guidance on Harmonisation of Requirements for Influenza Vaccines. For haemagglutination inhibition (HI), seroconversion is defined as achieving a post-vaccination titre of ≥ 40 for those participants with a pre-vaccination HI titre of < 10; significant increase is defined as a four-fold or greater increase in HI titre for those participants with a pre-vaccination HI titre of ≥ 10.
Time Frame: Approximately 21 days after vaccination
Population: The Evaluable Population comprised all participants who were vaccinated with the study vaccine, provided both pre- and post-vaccination antibody titre results, and were not excluded from the analyses (eg, for the use of a prohibited medication or a laboratory-confirmed influenza virus infection between Visits 1 and 2).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 60 | 58
percentage of participants
  A/Brisbane/59/2007 (H1N1) - like strain | 91.7 [81.6 to 97.2] | 53.4 [39.9 to 66.7]
  A/Brisbane/10/2007 (H3N2) - like strain | 93.3 [83.8 to 98.2] | 63.8 [50.1 to 76.0]
  B/Brisbane/60/2008 - like strain | 76.7 [64.0 to 86.6] | 46.6 [33.3 to 60.1]

2. Primary Outcome: The Geometric Mean Fold Increase (GMFI) in Antibody Titre After Vaccination.
Description: GMFI is defined as the geometric mean of the fold increases of post-vaccination antibody titre over the pre-vaccination antibody titre.
Time Frame: Approximately 21 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 60 | 58
percentage of participants
  A/Brisbane/59/2007 (H1N1) - like strain | 27.86 [19.339 to 40.129] | 5.02 [3.575 to 7.048]
  A/Brisbane/10/2007( H3N2) - like strain | 30.32 [21.003 to 43.772] | 9.80 [6.105 to 15.738]
  B/Brisbane/60/2008 - like strain | 12.85 [9.333 to 17.683] | 6.13 [4.121 to 9.107]

3. Primary Outcome: The Percentage of Evaluable Participants Achieving a HI Titre ≥ 40 or Single Radial Haemolysis (SRH) Area ≥ 25 mm2.
Time Frame: Approximately 21 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 60 | 58
percentage of participants
  A/Brisbane/59/2007 (H1N1) - like strain | 100.0 [94.0 to 100.0] | 91.4 [81.0 to 97.1]
  A/Brisbane/10/2007( H3N2) - like strain | 100.0 [94.0 to 100.0] | 94.8 [85.6 to 98.9]
  B/Brisbane/60/2008 - like strain | 85.0 [73.4 to 92.9] | 60.3 [46.6 to 73.0]

4. Secondary Outcome: The Frequency of Any Solicited Local Reactions.
Description: The number of participants reporting any solicited local reactions.
Time Frame: During the 4 days after vaccination (Day 0 plus 3 days)
Population: The Safety Population comprised all participants who received study vaccine.
Measure: Number; unit: participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 60 | 60
participants
  Any solicited local reaction | 32 | 22
  Any induration larger than 50 mm | 1 | 2
  Any erythema | 22 | 12
  Any pain | 26 | 14
  Any ecchymosis | 5 | 4

5. Secondary Outcome: The Frequency of Any Solicited Systemic Symptoms.
Description: The number of participants reporting any solicited systemic symptoms.
Time Frame: During the 4 days after vaccination (Day 0 plus 3 days)
Population: The Safety Population comprised all participants who received study vaccine.
Measure: Number; unit: participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 60 | 60
participants
  Any solicited systemic symptom | 7 | 5
  Any temperature above 38°C for 24 hours or longer | 1 | 0
  Any chills | 6 | 2
  Any malaise | 5 | 5

6. Secondary Outcome: The Incidence of Any Unsolicited Adverse Events (AEs).
Description: The number of participants reporting any unsolicited adverse events.
  Unsolicited adverse event (UAE) grading:
  Mild: Symptoms were easily tolerated and did not interfere with normal, everyday activities. Moderate: Enough discomfort to have caused some interference with normal, everyday activities. Severe: Symptoms that prevented normal, everyday activities.
Time Frame: After vaccination until the end of the study; approximately 21 days
Population: The Safety Population comprised all participants who received study vaccine.
Measure: Number; unit: participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 60 | 60
participants
  Number of participants with at least one UAE | 25 | 21
  Number of participants reporting mild UAE | 20 | 21
  Number of participants reporting moderate UAE | 12 | 3
  Number of participants reporting severe UAE | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 21 days after study vaccination for serious adverse events and unsolicited adverse events.
Description: The Safety Population comprised all participants who received study vaccine.
  Other adverse events presented were unsolicited adverse events up to approximately 21 days after study vaccination.
Arm/Group | Adults | Older Adults
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 14/60 | 11/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults (N=60) | Older Adults (N=60)
Injection site mass (General disorders) | 2 (2) | 3 (4)
Injection site erythema (General disorders) | 2 (2) | 3 (3)
Influenza like illness (General disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 8 (10) | 4 (5)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.